CLINICAL TRIAL: NCT03839823
Title: A Phase II Randomized Study of the Combination of Ribociclib Plus Goserelin Acetate With Hormonal Therapy Versus Physician Choice Chemotherapy in Premenopausal or Perimenopausal Patients With Hormone Receptor-positive/ HER2-negative Inoperable Locally Advanced or Metastatic Breast Cancer
Brief Title: Study to Compare the Combination of Ribociclib Plus Goserelin Acetate With Hormonal Therapy Versus Combination Chemotherapy in Premenopausal or Perimenopausal Patients With Advanced or Metastatic Breast Cancer
Acronym: RIGHT Choice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011A3201C
Record Dates: First submitted 2019-01-24; First posted 2019-02-15 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: HR-positive; HER2-negative; advanced breast cancer; Ribociclib; NSAI; Goserelin; Docetaxel / capecitabine; Paclitaxel/gemcitabine; Capecitabine/vinorelbine; CDK4/6 inhibitors; Phase II; ER-positive; PR-positive; Premenopausal; Perimenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Capecitabine; Vinorelbine; Paclitaxel; Gemcitabine; ribociclib; Letrozole; Anastrozole; Goserelin

STUDY DESIGN:
Intervention Model Description: This was a randomized, phase II, open label, multi-center trial comparing the combination of NSAI (letrozole or anastrozole) + goserelin + ribociclib versus combination chemotherapy (either of docetaxel/capecitabine or paclitaxel/gemcitabine or capecitabine/vinorelbine). Premenopausal or perimenopausal women with HR+, HER2- negative, advanced breast cancer with ECOG performance status of 0 to 2 and having symptomatic visceral metastases, or rapid progression of disease or impending visceral compromise, or markedly symptomatic non visceral disease were considered for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ribociclib 600 mg (Experimental): Combination of non-steroidal aromatase inhibitor: NSAI (letrozole or anastrozole) + goserelin + ribociclib.
  1. Ribociclib (600 mg) was dosed orally for the first 21 days out of a 28-day cycle.
  2. Letrozole (2.5 mg) or anastrozole (1 mg) were dosed orally daily (28 days out of the 28-day cycle).
  3. Goserelin (3.6 mg) was continuously released via a subcutaneous implant injected on Day 1 of each 28-day cycle (regardless of ribociclib treatment cycle) with an administration window of + 3 days.
  Interventions: Drug: Ribociclib; Drug: Letrozole OR Anastrozole; Drug: Goserelin
- Combination Chemotherapy (Active Comparator): Combination chemotherapies of docetaxel/capecitabine, paclitaxel/gemcitabine or capecitabine/vinorelbine were administered to patients enrolled in the control group. The chemotherapy regimen was decided by the treating physician.
  Interventions: Combination Product: Docetaxel / Capecitabine; Combination Product: Capecitabine / Vinorelbine; Combination Product: Paclitaxel / Gemcitabine

INTERVENTIONS:
Combination Product: Docetaxel / Capecitabine — Docetaxel (IV Infusion) / Capecitabine (Tablets for oral use):
  Docetaxel once, on day 1 of the 3-weeks cycle. Capecitabine twice daily, on Days 1 to 14, followed by a 1-week rest period, in 3 weeks cycle.
  Docetaxel (60 - 75 mg/m²)/capecitabine (1600 - 2500 mg/m²/day)
  Other Names: Combination chemotherapy group.; The chemotherapy regimen was decided by the treating physician.
  Arms: Combination Chemotherapy
Combination Product: Capecitabine / Vinorelbine — Capecitabine (Tablets for oral use) / Vinorelbine (Capsule for Oral use/IV infusion ).
  Capecitabine twice daily on day 1 to 14, followed by a 1-week rest period, in 3 weeks cycle.
  Vinorelbine, once, on Day 1 and Day 8 in 3 weeks cycles.
  Capecitabine (1600 - 2500 mg/m2/day)/vinorelbine (60 to 80 mg/m2/day [oral] or (25 to 30 mg/m2 [IV infusion]
  Other Names: Combination chemotherapy group.; The chemotherapy regimen was decided by the treating physician.
  Arms: Combination Chemotherapy
Combination Product: Paclitaxel / Gemcitabine — Paclitaxel (IV Infusion) / Gemcitabine (IV Infusion):
  Paclitaxel via 3-hour intravenous (IV) infusion on Day 1 in 3-weeks cycles, OR Paclitaxel via 1 hour intravenous (IV) infusion on Day 1 and day 8- in 3-weeks cycles.
  Gemcitabine at via 30 minute IV infusion on Day 1 and Day 8 in 3 weeks cycles.
  Paclitaxel (175 mg/m2) (on Day 1 in 3-weeks cycles)/ gemcitabine (1000 - 1250 mg/m2)
  OR
  Paclitaxel (80 - 90 mg/m2) (on Day 1 and Day 8 in 3-weeks cycles) / gemcitabine (800 - 1250 mg/m2)
  Other Names: Combination chemotherapy group.; The chemotherapy regimen was decided by the treating physician.
  Arms: Combination Chemotherapy
Drug: Ribociclib — Dose: 600 mg (200 mg * 3) Days 1 to 21 of each 28 day cycle Tablets for oral use
  Other Names: Endocrine treatment arm:; NSAI + goserelin+ ribociclib
  Arms: Ribociclib 600 mg
Drug: Letrozole OR Anastrozole — Letrozole:
  Dose: 2.5 mg All days of every cycle without interruption). Tablets for oral use
  Anastrozole:
  dose: 1 mg All days of every cycle without interruption. Tablets for oral use
  The NSAI (letrozole or anastrozole) will be decided by the treating physician.
  Other Names: Endocrine treatment arm:; NSAI + goserelin+ ribociclib
  Arms: Ribociclib 600 mg
Drug: Goserelin — Dose: 3.6 mg Day 1 of each 28 day cycle (regardless of ribociclib treatment cycle) with an administration window of + 3 days.
  Subcutaneous implant
  Other Names: Endocrine treatment arm:; NSAI + goserelin+ ribociclib
  Arms: Ribociclib 600 mg

SUMMARY:
To compare the combination of Ribociclib plus goserelin acetate with hormonal therapy versus combination chemotherapy in premenopausal or perimenopausal patients with advanced or metastatic breast cancer

DETAILED DESCRIPTION:
Patients were randomly assigned to one of the below treatment arms in 1:1 ratio:

* Ribociclib arm: non-steroidal aromatase inhibitor (NSAI) + goserelin + Ribociclib
* Combination chemotherapy arm: Either of docetaxel + capecitabine, paclitaxel + gemcitabine, or capecitabine + vinorelbine based chemotherapy treatment Randomization was stratified by (1) the presence of liver metastases (present or absent) (2) disease-free interval (DFI) < 2 years (yes or no, de novo stage 4 was defined as DFI > 2 years).

The study consisted of a 28-day Screening phase, treatment phase (including end of treatment (EOT) visit and safety follow-up), and survival follow-up. Patients received study treatment until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment for any other reason.

Patients were followed for survival regardless of treatment discontinuation for any reason (except if consent was withdrawn, patient was lost to follow-up, or until death) and regardless of achieving the primary endpoint, until death, withdrawal of consent, or loss to follow-up.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patient was an adult female ≥ 18 years old and < 60 years old at the time of informed consent.
2. Patient had a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer based on the most recently analyzed tissue sample and all tested by local laboratory. ER should have been more than 10% ER positive or Allred ≥5 by local laboratory testing.
3. Patient had HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1 + or 2 + If IHC is 2 +, a negative in situ hybridization (FISH, CISH, or SISH) test was required by local laboratory testing and based on the most recently analyzed tissue sample.
4. Women with inoperable locally advanced or metastatic breast cancer not amenable to curative therapy. Patients had to fulfill at least one of the following criteria to be considered that combination chemotherapy was needed according to PI's judgment. However, for patients who were eligible under inoperable locally advanced breast cancer or criteria 4c, the recruitment was stopped to enrich patient population with visceral metastases.

   * Symptomatic visceral metastases
   * Rapid progression of disease or impending visceral compromise.
   * Markedly symptomatic non-visceral disease if the treating physician opted to give chemotherapy for rapid palliation of patient's symptoms.
5. Patient was premenopausal or perimenopausal at the time of study entry.

   1. Premenopausal status was defined as either:

      * Patient had last menstrual period within the last 12 months. OR
      * If on tamoxifen within the past 14 days, plasma estradiol and FSH were in the premenopausal range, according to local laboratory definition.
      * In case of therapy induced amenorrhea, plasma estradiol and/or FSH were in the premenopausal range according to local laboratory definition.
      * Patients who had undergone bilateral oophorectomy were not eligible.
   2. Perimenopausal status was defined as neither premenopausal nor postmenopausal.
6. Patients had received neither prior hormonal therapy nor chemotherapy for advanced breast cancer, except LHRH agonist. Patients who received ≤ 14 days of tamoxifen or a NSAI (letrozole or anastrozole) with or without LHRH agonist for advanced breast cancer prior to randomization were eligible. Patient had measurable disease.

EXCLUSION CRITERIA;

1. Patient received prior systemic anti-cancer therapy (including hormonal therapy and chemotherapy, or any CDK4/6 inhibitor for advanced breast cancer).

   * Patients who received (neo) adjuvant therapy for breast cancer were eligible. If the prior neo (adjuvant) therapy included aromatase inhibitors, the treatment-free interval must have been greater than 12 months from the completion of aromatase inhibitor treatment until randomization.
   * If patients had disease recurrence during adjuvant tamoxifen treatment, disease-free interval (defined as duration between the date of patient received complete tumor resection for primary breast cancer lesion to the date of disease recurrence documented) must have been greater than 12 months.
   * Patients who were receiving ≤ 14 days of tamoxifen or NSAI or LHRH agonists ≤ 28 days for advanced breast cancer prior to randomization were eligible.
2. Patient had received extended-field radiotherapy ≤ 2 weeks prior to randomization or limited field radiotherapy ≤ 2 weeks prior to randomization, and had not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion). Patient from whom ≥ 25% of the bone marrow had been previously irradiated were also excluded.
3. Patient had a concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated, basal or squamous cell skin carcinoma or curatively resected cervical cancer in situ.
4. Patients who had lung metastases with oxygen demand in resting status.
5. Patients who had liver metastases with bilirubin > 1.5 ULN.
6. Patients with CNS involvement unless they met ALL of the following criteria:

   * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment.
   * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases.
   * Leptomeningeal metastases was not allowed, even with stable clinical condition.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patient was an adult female ≥ 18 years old and < 60 years old at the time of informed consent.
Enrollment: 222 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- Egypt (2):
  - Novartis Investigative Site, Cairo
  - Novartis Investigative Site, Giza
- India (6):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Amman, Jordan
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Saida
  - Novartis Investigative Site, Tripoli
- Malaysia (5):
  - Novartis Investigative Site, Johor Bahru, Johor
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Pulau Pinang
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Pushkin Saint Petersburg
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- South Africa (2):
  - Novartis Investigative Site, Durban, KwaZulu-Natal
  - Novartis Investigative Site, Pretoria
- Taiwan (5):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Cankaya Ankara, Turkey
  - Novartis Investigative Site, Kecioren Ankara, Turkey
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Malatya
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Lu YS, Mahidin EIBM, Azim H, Eralp Y, Yap YS, Im SA, Rihani J, Gokmen E, El Bastawisy A, Karadurmus N, Lim YN, Lim CS, Duc LT, Chung WP, Babu KG, Penkov K, Bowles J, Alfaro TD, Wu J, Gao M, Slimane K, El Saghir NS. Final Results of RIGHT Choice: Ribociclib Plus Endocrine Therapy Versus Combination Chemotherapy in Premenopausal Women With Clinically Aggressive Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer. J Clin Oncol. 2024 Aug 10;42(23):2812-2821. doi: 10.1200/JCO.24.00144. Epub 2024 May 21. PMID 38771995
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2079

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Started | 112 | 110
Treated | 112 | 100
Not Treated | 0 | 10
Completed | 35 | 17
Not Completed | 77 | 93
Not completed — Adverse Event | 8 | 4
Not completed — Death | 1 | 0
Not completed — Physician Decision | 1 | 5
Not completed — Progressive Disease (PD) | 65 | 65
Not completed — Subject Decision | 2 | 9
Not completed — Not Treated | 0 | 10

BASELINE CHARACTERISTICS:
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy | Total
Number analyzed (Participants) | 112 | 110 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (6.26) | 42.0 (6.72) | 42.5 (6.49)
Sex/Gender, Customized [Number; unit: participants]
  Female | 112 | 110 | 222
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 60 | 58 | 118
  White | 51 | 52 | 103
  Black or African American | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 108 | 108 | 216
  Not Reported | 3 | 1 | 4
  Hispanic or Latino | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: cm] — Population: Data are reported for participants in the full analysis set who had available data.
  cm
    number analyzed (Participants) | 111 | 109 | 220
    (all) | 157.50 (7.489) | 158.34 (6.548) | 157.92 (7.035)

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the date of randomization to the date of the first documented progression as per local review and according to RECIST 1.1 or death due to any cause. PFS was censored at the date of the last adequate tumor assessment if no PFS event was observed at the time of last patient, last visit (LPLV).
Time Frame: Up to approximately 34 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
months | 21.8 [17.4 to 26.7] | 12.8 [10.1 to 18.4]
Statistical Analysis 1: Comparison: Ribociclib 600 mg vs Combination Chemotherapy; Test type: Superiority; p = 0.003, one-sided stratified logrank test; Hazard Ratio (HR) = 0.611, 95% CI 2-sided [0.429 to 0.870]

2. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from the date of randomization/start of treatment to the earliest of date of progression, date of death due to any cause, change to other anti-cancer therapy, or date of discontinuation due to reasons other than 'Protocol violation' or 'Administrative problems'. Patients who did not achieve a confirmed PR or CR were censored at: the maximum follow-up time (i.e., LPLV - first patient first visit [FPFV] used for the analysis) for patients who had a PFS event (i.e., either progressed or died due to any cause); the last adequate tumor assessment date for all other patients.
Time Frame: Up to approximately 34 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
months | 18.6 [13.2 to 24.0] | 9.1 [7.6 to 12.3]
Statistical Analysis 1: Comparison: Ribociclib 600 mg vs Combination Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.497, 95% CI [0.363 to 0.680]

3. Secondary Outcome: 3-month Treatment Failure Rate
Description: Treatment failure rate was defined as the percentage of patients who discontinued the study treatment due to progressive disease, death due to any cause, change to other anti-cancer therapy, or discontinuation due to reasons other than protocol violation or administrative problems.
Time Frame: Up to approximately 3 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
percentage of participants | 11.6 [6.3 to 19.0] | 21.8 [14.5 to 30.7]
Statistical Analysis 1: Comparison: Ribociclib 600 mg vs Combination Chemotherapy; Test type: Superiority; p = 0.020, Cochran-Mantel-Haenszel

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) was defined as the percentage of patients with a best overall response (BOR) of complete response (CR) or partial response (PR, response without image confirmation), as per local review and according to RECIST 1.1.
Time Frame: Up to approximately 34 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
percentage of participants | 66.1 [56.5 to 74.7] | 61.8 [52.1 to 70.9]
Statistical Analysis 1: Comparison: Ribociclib 600 mg vs Combination Chemotherapy; Test type: Superiority; p = 0.255, Cochran-Mantel-Haenszel

5. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate was defined as the percentage of patients with a BOR of CR, PR, or stable disease (SD, response without image confirmation) lasting 24 weeks or longer, as defined by RECIST 1.1.
Time Frame: Up to approximately 34 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
percentage of participants | 81.3 [72.8 to 88.0] | 74.5 [65.4 to 82.4]
Statistical Analysis 1: Comparison: Ribociclib 600 mg vs Combination Chemotherapy; Test type: Superiority; p = 0.116, Cochran-Mantel-Haenszel

6. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from the date of randomization to the first documented response of either CR or PR, which must be subsequently confirmed, as defined by RECIST 1.1. Patients who did not achieve a confirmed PR or CR were censored at: the maximum follow-up time (i.e., LPLV - FPFV used for the analysis) for patients who had a PFS event (i.e., either progressed or died due to any cause); the last adequate tumor assessment date for all other patients.
Time Frame: Up to approximately 34 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
months | 4.9 [4.5 to 8.3] | 3.2 [2.7 to 4.7]
Statistical Analysis 1: Comparison: Ribociclib 600 mg vs Combination Chemotherapy; Test type: Superiority; Hazard Ratio (HR) = 0.762, 95% CI 2-sided [0.546 to 1.064]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause. If a patient was not known to have died at the time of LPLV, then OS was censored at the last contact date.
Time Frame: Up to approximately 46 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
months | NA [38.6 to NA] — Median and the upper limit of 95% CI were not estimable due to an insufficient number of participants with events. | NA [30.8 to NA] — Median and the upper limit of 95% CI were not estimable due to an insufficient number of participants with events.

8. Secondary Outcome: Change From Baseline in the Global Health Status/Quality of Life (QOL) Scale Score by Using the Functional Assessment of Cancer Therapy - Breast (FACT-B) Questionnaire
Description: FACT-B is a self-reported instrument that measures multidimensional quality of life (QOL) in patients with breast cancer. The FACT-B consists of 37 questions that address physical, social, emotional, and functional well-being, with specific questions relevant to women with breast cancer. Each item has a score range of 0 (Not at all) to 4 (Very much), with a total score ranging from 0-148. The higher the score, the better the QOL reported by the participant. A positive change from baseline indicates improvement in QoL.
Time Frame: Up to approximately 46 months
Population: The full analysis set comprised all patients to whom study treatment was assigned by randomization. Results are reported for participants with data available at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 110
score on a scale
  Week 6 n=109,90: number analyzed (Participants) | 109 | 90
  Week 6 n=109,90 | 4.3 (13.45) | 4.8 (15.33)
  Week 12 n=100,82: number analyzed (Participants) | 100 | 82
  Week 12 n=100,82 | 5.5 (16.28) | 4.4 (16.73)
  Week 20 n=94,76: number analyzed (Participants) | 94 | 76
  Week 20 n=94,76 | 5.9 (18.18) | 4.9 (17.51)
  Week 28 n=87,67: number analyzed (Participants) | 87 | 67
  Week 28 n=87,67 | 7.9 (17.54) | 6.2 (16.15)
  Week 36 n=79,56: number analyzed (Participants) | 79 | 56
  Week 36 n=79,56 | 7.3 (18.65) | 6.5 (16.60)
  Week 44 n=75,50: number analyzed (Participants) | 75 | 50
  Week 44 n=75,50 | 7.2 (18.33) | 6.6 (14.39)
  Week 56 n=68,38: number analyzed (Participants) | 68 | 38
  Week 56 n=68,38 | 7.3 (20.79) | 4.7 (16.13)
  Week 68 n=64,32: number analyzed (Participants) | 64 | 32
  Week 68 n=64,32 | 7.4 (19.86) | 5.1 (16.92)
  Week 80 n=53,22: number analyzed (Participants) | 53 | 22
  Week 80 n=53,22 | 7.1 (25.49) | 7.0 (14.50)
  Week 92 n=45,16: number analyzed (Participants) | 45 | 16
  Week 92 n=45,16 | 9.4 (22.46) | 9.6 (20.24)
  Week 104 n=36,12: number analyzed (Participants) | 36 | 12
  Week 104 n=36,12 | 7.9 (22.26) | 15.1 (13.04)
  Week 116 n=29,8: number analyzed (Participants) | 29 | 8
  Week 116 n=29,8 | 5.3 (23.58) | 15.8 (7.92)
  Week 128 n=26,8: number analyzed (Participants) | 26 | 8
  Week 128 n=26,8 | 2.8 (24.17) | 17.0 (11.40)
  Week 140 n=21,6: number analyzed (Participants) | 21 | 6
  Week 140 n=21,6 | 10.9 (24.30) | 20.8 (13.80)
  Week 152 n=17,5: number analyzed (Participants) | 17 | 5
  Week 152 n=17,5 | 3.6 (20.39) | 17.0 (14.06)
  Week 164 n=10,1: number analyzed (Participants) | 10 | 1
  Week 164 n=10,1 | 1.6 (16.56) | 33.8 (NA) — Due to a single participant at this timepoint, standard deviation was not applicable.
  Week 176 n=3,1: number analyzed (Participants) | 3 | 1
  Week 176 n=3,1 | 16.9 (31.39) | 39.7 (NA) — Due to a single participant at this timepoint, standard deviation was not applicable.
  Week 188 n=1,0: number analyzed (Participants) | 1 | 0
  Week 188 n=1,0 | 7.0 (NA) — Due to a single participant at this timepoint, standard deviation was not applicable. |

9. Secondary Outcome: Number of Patients With Adverse Events, Categorized by Severity
Description: Adverse events were assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 or higher. If CTCAE grading did not exist for an adverse event, the severity of mild, moderate, severe, and life-threatening, corresponding to Grades 1 - 4, were used. A patient with multiple severity grades for an AE was only counted under the maximum grade. Data for Grades 3 and 4 are reported.
Time Frame: Up to approximately 46 months
Population: The safety set included all patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 100
Participants
  All grades | 112 | 100
  Grade 3 | 71 | 62
  Grade 4 | 18 | 11

10. Secondary Outcome: Number of Patients With Laboratory Abnormalities
Description: Grading of laboratory values was assigned programmatically as per NCI Common Terminology Criteria for Adverse Events (CTCAE) version available at the time of analysis. The calculation of CTCAE grades was based on the observed laboratory values only, clinical assessments were not be taken into account. CTCAE Grade 0 was assigned for all non-missing values not graded as 1 or higher. Grade 5 was not used. For laboratory tests where grades were not defined by CTCAE available at the time of analysis, results were categorized as low/normal/high based on laboratory normal ranges.
Time Frame: Up to approximately 46 months
Population: The safety set included all patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 100
Participants
  Hemoglobin - Hypo: Grades 1/2 | 82 | 73
  Hemoglobin - Hypo: Grade 3 | 5 | 11
  Hemoglobin - Hypo: Grade 4 | 0 | 0
  Leukocytes - Hypo: Grades 1/2 | 71 | 54
  Leukocytes - Hypo: Grade 3 | 34 | 8
  Leukocytes - Hypo: Grade 4 | 0 | 1
  Lymphocytes (absolute) - Hyper: Grades 1/2 | 3 | 10
  Lymphocytes (absolute) - Hyper: Grade 3 | 0 | 0
  Lymphocytes (absolute) - Hyper: Grade 4 | 0 | 0
  Lymphocytes (absolute) - Hypo: Grades 1/2 | 55 | 37
  Lymphocytes (absolute) - Hypo: Grade 3 | 21 | 3
  Lymphocytes (absolute) - Hypo: Grade 4 | 1 | 4
  Neutrophils (absolute) - Hypo: Grades 1/2 | 40 | 35
  Neutrophils (absolute) - Hypo: Grade 3 | 55 | 23
  Neutrophils (absolute) - Hypo: Grade 4 | 10 | 9
  Platelets - Hypo: Grades 1/2 | 37 | 27
  Platelets - Hypo: Grade 3 | 2 | 2
  Platelets - Hypo: Grade 4 | 1 | 1
  Prothrombin Intl. Normalized Ratio - Hyper: Grades 1/2 | 0 | 8
  Prothrombin Intl. Normalized Ratio - Hyper: Grade 3 | 0 | 0
  Prothrombin Intl. Normalized Ratio - Hyper: Grade 4 | 0 | 0

11. Secondary Outcome: Post-Hoc: All Collected Deaths
Description: On-treatment deaths due to any cause were collected from first dose of study medication to 30 days after the last dose of study treatment. Post-treatment survival follow-up deaths were collected from day 31 after last dose of study medication to end of study.
Time Frame: On-treatment deaths: Up to approximately 46 months. Post-treatment survival follow-up deaths: Up to approximately 2 additional months.
Population: All participants to whom study treatment was assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Ribociclib 600 mg | Combination Chemotherapy
Number analyzed (Participants) | 112 | 100
Participants
  On-treatment deaths | 5 | 0
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 107 | 92
  Post-treatment survival follow-up deaths | 29 | 29
  All deaths | 34 | 29

ADVERSE EVENTS:
Time Frame: From day of first dose of study medication to last dose of study medication plus 30 days, up to approximately 46 months. Deaths were collected in the post treatment survival follow-up from 31 days after last dose of study medication until the end of the study, up to approximately 2 additional months. These were not considered AEs.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. Deaths in the post-treatment survival follow-up were not considered adverse events. The total number at risk in the post-treatment survival includes patients that entered the post-treatment survival follow-up period.
Groups:
- Ribociclib 600 mg (On-treatment); Combination Chemotherapy (On-treatment): AEs during the on-treatment period (up to 30 days post-treatment)
- Ribociclib 600 mg (Post-treatment Survival Follow-up); Combination Chemotherapy (Post-treatment Survival Follow-up): Deaths collected in the post-treatment survival follow-up period (starting from Day 31 post-treatment). No AEs were collected during this period.
Arm/Group | Ribociclib 600 mg (On-treatment) | Combination Chemotherapy (On-treatment) | Ribociclib 600 mg (Post-treatment Survival Follow-up) | Combination Chemotherapy (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 5/112 | 0/100 | 29/107 | 29/92
Serious Adverse Events (participants affected / at risk) | 17/112 | 16/100 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 112/112 | 100/100 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib 600 mg (On-treatment) (N=112) | Combination Chemotherapy (On-treatment) (N=100) | Ribociclib 600 mg (Post-treatment Survival Follow-up) (N=0) | Combination Chemotherapy (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | NA | NA
Angina pectoris (Cardiac disorders) | 1 | 0 | NA | NA
Cardiac tamponade (Cardiac disorders) | 0 | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | NA | NA
Disease progression (General disorders) | 1 | 0 | NA | NA
Localised oedema (General disorders) | 0 | 1 | NA | NA
Non-cardiac chest pain (General disorders) | 1 | 0 | NA | NA
Pyrexia (General disorders) | 1 | 0 | NA | NA
Abdominal sepsis (Infections and infestations) | 1 | 0 | NA | NA
COVID-19 (Infections and infestations) | 4 | 0 | NA | NA
Catheter site cellulitis (Infections and infestations) | 0 | 1 | NA | NA
Dengue fever (Infections and infestations) | 0 | 1 | NA | NA
Herpes zoster (Infections and infestations) | 0 | 1 | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | NA | NA
Peritonitis bacterial (Infections and infestations) | 0 | 1 | NA | NA
Pneumonia (Infections and infestations) | 2 | 2 | NA | NA
Sepsis (Infections and infestations) | 2 | 0 | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 1 | NA | NA
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | NA | NA
Electrocardiogram T wave inversion (Investigations) | 1 | 0 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | NA | NA
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | NA | NA
Menopause (Social circumstances) | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ribociclib 600 mg (On-treatment) (N=112) | Combination Chemotherapy (On-treatment) (N=100) | Ribociclib 600 mg (Post-treatment Survival Follow-up) (N=0) | Combination Chemotherapy (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 40 | 42 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 29 | 14 | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 11 | 6 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 73 | 38 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 7 | NA | NA
Constipation (Gastrointestinal disorders) | 16 | 12 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 3 | 26 | NA | NA
Nausea (Gastrointestinal disorders) | 14 | 27 | NA | NA
Stomatitis (Gastrointestinal disorders) | 3 | 7 | NA | NA
Vomiting (Gastrointestinal disorders) | 7 | 30 | NA | NA
Fatigue (General disorders) | 9 | 25 | NA | NA
Oedema peripheral (General disorders) | 2 | 9 | NA | NA
Pyrexia (General disorders) | 6 | 16 | NA | NA
COVID-19 (Infections and infestations) | 17 | 10 | NA | NA
Cellulitis (Infections and infestations) | 2 | 7 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 8 | 4 | NA | NA
Alanine aminotransferase increased (Investigations) | 23 | 30 | NA | NA
Aspartate aminotransferase increased (Investigations) | 23 | 29 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 12 | 8 | NA | NA
Blood bilirubin increased (Investigations) | 6 | 1 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 7 | 11 | NA | NA
Electrocardiogram QT prolonged (Investigations) | 23 | 11 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 18 | 8 | NA | NA
Lipase increased (Investigations) | 7 | 2 | NA | NA
Lymphocyte count decreased (Investigations) | 8 | 3 | NA | NA
Neutrophil count decreased (Investigations) | 28 | 16 | NA | NA
White blood cell count decreased (Investigations) | 27 | 12 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | 8 | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 7 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 7 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 7 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 13 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 11 | NA | NA
Dizziness (Nervous system disorders) | 7 | 6 | NA | NA
Headache (Nervous system disorders) | 8 | 6 | NA | NA
Neuropathy peripheral (Nervous system disorders) | 3 | 14 | NA | NA
Insomnia (Psychiatric disorders) | 9 | 6 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 12 | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 20 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 5 | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 32 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 7 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 10 | 7 | NA | NA
Hot flush (Vascular disorders) | 12 | 0 | NA | NA
Hypertension (Vascular disorders) | 9 | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT03839823/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03839823/SAP_001.pdf